CLINICAL TRIAL: NCT04576429
Title: Immune Profiles Evolution in Patients Treated by Immunotherapy for Melanoma
Brief Title: Immune Profiles Evolution Under Immunotherapy for Melanoma
Acronym: EPITHEM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200947; 2019-A02695-52 (Registry Identifier: IDRCB)
Record Dates: First submitted 2020-09-14; First posted 2020-10-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Melanoma
Keywords: melanoma; immunotherapy; immune profiles
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Procedure: venous puncture; Procedure: tumoral biopsy
- comparator group (Active Comparator)
  Interventions: Procedure: venous puncture; Procedure: tumoral biopsy

INTERVENTIONS:
Procedure: venous puncture — Venous punctures will be performed:
  for patients of cohort A and B1:
  * before the first immune checkpoint inhibitors monoclonal antibodies infusion (baseline);
  * between week 6 and week 8 (before the immune checkpoint inhibitors monoclonal antibodies infusion);
  * each 3 months up to 12 months.
  for patients of cohort B2:
  * before the radiotherapy;
  * within the 6 weeks after the end of radiotherapy;
  * at the 2 following evaluations (every 3 months).
Procedure: tumoral biopsy — Cutaneous biopsy: superficial skin, or extended skin biopsy, if it is indicated for patient's care.

SUMMARY:
The primary objective of the study aims to compare the immune profiles (circulating cytokines and lymphocytes) before and after (6 to 8 weeks) the first infusion of immune checkpoint inhibitors in patients with melanoma treated in the adjuvant setting(cohort A) or in metastatic setting(cohort B); and to study the association of these immune profiles with relapse- or progression-free survival.

DETAILED DESCRIPTION:
This study will analyse the association of biomarkers with relapse- or progression-free survival of stage III or IV melanoma patients, divided in 3 sub-cohorts:

* Patients treated in the adjuvant setting (cohort A): new user of immune checkpoint blockers.
* Patients treated in the metastatic setting (cohort B): - B1: new users of immune checkpoint blockers; - B2: prevalent users of immune checkpoint blockers treated with complementary radiotherapy.

For patients of cohort A and B1, immune profiles characteristics will be evaluated before initiation of treatment (=baseline), and at each radiological evaluation of the tumour response, up to maximum 12 months as duration.

The maximal duration of treatment will be 12 months for patients treated in the adjuvant setting. For metastatic patients, the duration of treatment will be decided by physician according to different factors (responses, progression, toxicities, ...).

For patients in cohort B2, the characteristics of the immune profiles will be evaluated before radiotherapy initiation,, within 6 weeks after the end of radiotherapy, then at the 2 following radiological evaluations of the tumour response

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years;
* Totally resected stage III or IV melanoma totally resected, treated with a immune therapy (pembrolizumab or nivolumab ou other immune checkpoint inhibitors) as adjuvant treatment;
* Unresectable stage IIIC/D or IV metastatic melanoma, treated with immune therapy (pembrolizumab or nivolumab or immune checkpoint inhibitors) which should be associated by a radiotherapy ;
* Patient has been informed about the study and signed the consent;
* Affiliated to the French social security scheme.

Exclusion Criteria:

* Pregnant or breastfeeding woman;
* Patient refusal;
* Patient receiving a immunosuppressor;
* Undergo a general corticotherapy of > 10 mg/kg/day since more than 7 days;
* Patient who participate to another blind interventional study receiving blinded treatment;
* Patient without any social protection by organization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Rate of relapse/progression-free survival | at 5 years
  Will be noted: all progression and event of death. Survival rate will be calculated between the event's day and the beginning of anticancer treatment.

SECONDARY OUTCOMES:
immunity profiles | quarterly up to 12 months
  ELISA Multiplex method will be used to analyse inflammatory human cytokines in plasma. This method will performe an assay 45-plex fixed panel :
  Analytes Included in the Assay
  * CCL2/JE/MCP-1
  * CCL3/MIP-1 alpha
  * CCL4/MIP-1 beta
  * CCL5/RANTES
  * CCL11/Eotaxin
  * CCL19/MIP-3 beta
  * CCL20/MIP-3 alpha
  * CD40 Ligand/TNFSF5
  * CX3CL1/Fractalkine
  * CXCL1/GRO alpha/KC/CINC-1
  * CXCL2/GRO beta/MIP-2/CINC-3
  * CXCL10/IP-10/CRG-2
  * EGF
  * FGF basic/FGF2/bFGF
  * Flt-3 Ligand/FLT3L
  * G-CSF
  * GM-CSF
  * Granzyme B
  * IFN-alpha 2/IFNA2
  * IFN-beta
  * IFN-gamma
  * IL-1 alpha/IL-1F1
  * IL-1 beta/IL-1F2
  * IL-1ra/IL-1F3
  * IL-2
  * IL-3
  * IL-4
  * IL-5
  * IL-6
  * IL-7
  * IL-8/CXCL8
  * IL-10
  * IL-12 p70
  * IL-13
  * IL-15
  * IL-17/IL-17A
  * IL-17E/IL-25
  * IL-33
  * PD-L1/B7-H1
  * PDGF-AA
  * PDGF-AB/BB
  * TGF-alpha
  * TNF-alpha
  * TRAIL/TNFSF10
  * VEGF

CONTACTS AND LOCATIONS:
Overall Officials: Elisa FUNCK-BRENTANO, MD, Principal Investigator — Dermato-oncology department, Ambroise Paré hospital, APHP; Jean-François EMILE, MD, PhD, Study Director — Pathology department, Ambroise Paré hospital, APHP
Locations (1):
- Dermato-oncology department, Ambroise Paré hospital, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No